CLINICAL TRIAL: NCT04573660
Title: Abbott Vascular Medical Device Registry
Acronym: AV-MDR
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10349
Record Dates: First submitted 2020-09-23; First posted 2020-10-05 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Acute Myocardial Infarction; Restenoses, Coronary; Coronary Artery Lesions; Venous Embolism; Arterial Embolism
Keywords: Coronary and peripheral stents; ABT-CIP-10349; Vascular plugs; Pacing catheters; Measurement and imaging (FFR and OCT); Peripheral dilatation catheters; Coronary dilatation catheters; Coronary and peripheral guidewires; Vessel closure/compression devices; Vascular access introducers
MeSH Terms: conditions — Coronary Restenosis; Ornithine Carbamoyltransferase Deficiency Disease | interventions — Weights and Measures; Diagnostic Imaging; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (9):
- Coronary and peripheral stents: Participants in the Coronary and peripheral stents arm will receive Coronary and peripheral stents
  Interventions: Device: Coronary and peripheral stents
- Pacing catheters: Participants in the Pacing catheters arm will receive Pacing catheters
  Interventions: Device: Pacing catheters
- Vascular plugs: Participants in the Vascular plugs arm will receive Vascular plugs
  Interventions: Device: Vascular plugs
- Measurement and imaging (FFR and OCT): Participants in the Measurement and imaging (FFR and OCT) arm will receive Measurement and imaging (FFR and OCT)
  Interventions: Device: Measurement and imaging (FFR and OCT)
- Peripheral dilatation catheters: Participants in the Peripheral dilatation catheters arm will receive Peripheral dilatation catheters
  Interventions: Device: Peripheral dilatation catheters
- Coronary dilatation catheters: Participants in the Coronary dilatation catheters arm will receive Coronary dilatation catheters
  Interventions: Device: Coronary dilatation catheters
- Coronary and peripheral guidewires: Participants in the Coronary and peripheral guidewires arm will receive Coronary and peripheral guidewires
  Interventions: Device: Coronary and peripheral guidewires
- Vessel closure/compression devices: Participants in the Vessel closure/compression devices arm will receive Vessel closure/compression devices
  Interventions: Device: Vessel closure/compression devices
- Vascular access introducers: Participants in the Vascular access introducers devices arm will receive Vascular access introducers
  Interventions: Device: Vascular access introducers

INTERVENTIONS:
Device: Coronary and peripheral stents — The participants in the Coronary and peripheral stents arm will receive Coronary and peripheral stents
  Groups: Coronary and peripheral stents
Device: Pacing catheters — The participants in the Pacing catheters arm will receive Pacing catheters
  Groups: Pacing catheters
Device: Vascular plugs — The participants in the Vascular plugs arm will receive Vascular plugs
  Groups: Vascular plugs
Device: Measurement and imaging (FFR and OCT) — The participants in the Measurement and imaging (FFR and OCT) arm will receive Measurement and imaging (FFR and OCT)
  Groups: Measurement and imaging (FFR and OCT)
Device: Peripheral dilatation catheters — The participants in the Peripheral dilatation catheters will receive Peripheral dilatation catheters
  Groups: Peripheral dilatation catheters
Device: Coronary dilatation catheters — The participants in the Coronary dilatation catheters will receive Coronary dilatation catheters
  Groups: Coronary dilatation catheters
Device: Coronary and peripheral guidewires — The participants in the Coronary and peripheral guidewires will receive Coronary and peripheral guidewires
  Groups: Coronary and peripheral guidewires
Device: Vessel closure/compression devices — The participants in the Vessel closure/compression devices will receive Vessel closure/compression devices
  Groups: Vessel closure/compression devices
Device: Vascular access introducers — The participants in the Vascular access introducers arm will receive Vascular access introducers
  Groups: Vascular access introducers

SUMMARY:
The AV-MDR is a prospective, non-randomized, open-label, multi-center registry. The purpose of the AV-MDR study is to proactively collect and evaluate clinical data on the usage of the devices in scope within their intended use with the aim of confirming safety and performance throughout their expected lifetime, ensuring the continued acceptability of identified risks, detecting emerging risks on the basis of factual evidence, ensuring the continued acceptability of the benefit-risk ratio, and identifying possible systematic misuse or off-label usage such that the intended use can be verified as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age.
2. Subject has a planned procedure, or underwent a procedure, that will use/used one or more Abbott target devices covered in this registry.
3. Subject is willing and able to comply with, or has already completed, the follow-up schedule specified in this protocol.
4. Subject must provide written informed consent prior to any clinical investigation-related data collection or be enrolled under an IRB/EC approved waiver of consent.

Exclusion Criteria:

1. Subject has active symptoms and/or a positive test result of COVID-19 or other rapidly spreading novel infectious agent within the prior 2 months of the date of procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll subjects 18 years and older of all genders in which at least one Abbott target device specified in the CIP is used. Outcomes will be collected on any ancillary devices in scope, but patients will not be enrolled for use of an ancillary device without treatment with any target device. Patients must meet all general eligibility criteria and provide written informed consent or be enrolled under an IRB/EC approved waiver of consent, prior to sites' collection of patient data for the investigation.
Sampling Method: Non-Probability Sample
Enrollment: 3784 (Estimated)
Dates: Start 2020-10-25 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Coronary Stents - Number of participants with composite of all-cause death, MI or target lesion revascularization (TLR) | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Composite of all-cause death, MI or target lesion revascularization (TLR) will be assessed among the patients who receive Coronary Stents.
Coronary Stents - Number of participants with composite of all-cause death, MI or target lesion revascularization (TLR) | 30 days
  Composite of all-cause death, MI or target lesion revascularization (TLR) will be assessed among the patients who receive Coronary Stents.
Coronary Stents - Number of participants with composite of all-cause death, MI or target lesion revascularization (TLR) | 12 months
  Composite of all-cause death, MI or target lesion revascularization (TLR) will be assessed among the patients who receive Coronary Stents.
Peripheral Stents - Number of participants with composite of all-cause death, amputation, and TLR | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Composite of all-cause death, amputation, and TLR will be assessed among the patients who receive Peripheral Stents.
Peripheral Stents - Number of participants with composite of all-cause death, amputation, and TLR | 30 days
  Composite of all-cause death, amputation, and TLR will be assessed among the patients who receive Peripheral Stents.
Peripheral Stents - Number of participants with composite of all-cause death, amputation, and TLR | 12 months
  Composite of all-cause death, amputation, and TLR will be assessed among the patients who receive Peripheral Stents.
Peripheral Stents (Renal Indication) - Number of participants with composite of all-cause death, ipsilateral nephrectomy, Embolic events resulting in kidney damage or TLR | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Composite of all-cause death, ipsilateral nephrectomy, Embolic events resulting in kidney damage or TLR will be assessed among the patients who receive Peripheral Stents (Renal Indication).
Peripheral Stents (Renal Indication) - Number of participants with composite of all-cause death, ipsilateral nephrectomy, Embolic events resulting in kidney damage or TLR | 30 days
  Composite of all-cause death, ipsilateral nephrectomy, Embolic events resulting in kidney damage or TLR will be assessed among the patients who receive Peripheral Stents (Renal Indication).
Peripheral Stents (Renal Indication) - Number of participants with composite of TLR | 12 months
  Composite of TLR will be assessed among the patients who receive Peripheral Stents (Renal Indication).
Pacing Catheters - Number of participants with composite of potential complications (venous thrombosis, pulmonary emboli, arrhythmias, perforation) | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Composite of potential complications (venous thrombosis, pulmonary emboli, arrhythmias, perforation) will be assessed among the patients who receive Pacing Catheters.
Pacing Catheters - Loss of capture (assessed based on physiological parameter-ECG) | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Loss of capture (average time of loss of capture across patients) will be assessed among the patients who receive Pacing Catheters. ECG is used to measure whether the pacing device stimulates the heart. Absence of a stimulation is considered a loss of capture.
Vascular Plugs - Number of participants with composite of potential complications (Implant success, occlusion success, migration) | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Composite of potential complications including implant success, occlusion success, migration will be assessed among the patients who receive Vascular Plugs.
Vascular Plugs - Number of participants with composite of occlusion success and migration | 30 days
  Composite of occlusion success and migration will be assessed among the patients who receive Vascular Plugs.
Fractional flow reserve - Number of participants with composite of vessel dissection, perforation, and thromboembolism | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Composite of vessel dissection, perforation, and thromboembolism during procedure will be assessed among the patients who receive Fractional flow reserve (FFR).
Fractional flow reserve - Number of participants with signal drift (Signal drift between measurements (Pd/Pa** pressure drift >0.03; <0.97 or >1.03) | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Signal drift (Signal drift between measurements (Pd/Pa** pressure drift >0.03; <0.97 or >1.03) will be assessed among the patients who receive FFR.
Optical Coherence Tomography Products - Number of participants with Intraprocedural complications (number of dissections ≥type B, slow flow or no reflow, thrombus, abrupt closure, perforation) | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Intraprocedural complications will be assessed among the patients who receive Optical Coherence Tomography (OCT).
Optical Coherence Tomography Products - Number of participants with Successful crossing and image quality pre-PCI | During procedure - Before the stent is implanted (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Successful crossing and image quality pre- PCI will be assessed among the patients who receive OCT.
Optical Coherence Tomography Products - Number of participants with Successful crossing and image quality post-PCI | During procedure - Between 10-30 minutes post-PCI (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Successful crossing and image quality post-PCI will be assessed among the patients who receive OCT.
Peripheral Dilatation Catheters - Number of participants with Composite of major adverse events | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Composite of major adverse events (e.g., distal embolization, dissection, perforation, amputation primary to balloon usage, total occlusion, abrupt closure, renal failure primary to balloon usage will be assessed among the patients who receive Peripheral Dilatation Catheters.
Peripheral Dilatation Catheters - Number of participants with Device success (Successful delivery, Successful inflation, Successful deflation, Successful withdrawal) (assessed based on physiological parameters) | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Device success (Successful delivery, Successful inflation, Successful deflation, Successful withdrawal) will be assessed among the patients who receive Peripheral Dilatation Catheters. Device success can be summarized as the successful treatment with the device.
Coronary Guidewires - Number of participants with Composite of major adverse events | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Composite of major adverse events (e.g., vessel perforation, dissection, occlusion, embolism) will be assessed among the patients who receive Coronary Guidewires.
Coronary Guidewires - Number of participants with Device success (Successfully placed, Successfully introduce/position diagnostic/interventional device, Successfully reach/cross target lesion) (assessed based on physiological parameters) | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Device success (Successfully placed, Successfully introduce/position diagnostic/interventional device, Successfully reach/cross target lesion will be assessed among the patients who receive Coronary Guidewires. Device success can be summarized as the successful treatment with the device.
Peripheral Guidewires - Number of participants with Composite of major adverse events | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Composite of major adverse events (e.g., vessel perforation, dissection, occlusion, embolism) will be assessed among the patients who receive Peripheral Guidewires.
Peripheral Guidewires - Number of participants with Device success (Successfully placed, Successfully introduce/position diagnostic/interventional device, Successfully reach/cross target lesion) (assessed based on physiological parameters) | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Device success (Successfully placed, Successfully introduce/position diagnostic/interventional device, Successfully reach/cross target lesion will be assessed among the patients who receive Peripheral Guidewires. Device success can be summarized as the successful treatment with the device.
Coronary Dilatation Catheters - Number of participants with Composite of major adverse events | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Composite of major adverse events (e.g., distal embolization, dissection, perforation, amputation primary to balloon usage, total occlusion, abrupt closure, renal failure primary to balloon usage will be assessed among the patients who receive Coronary Dilatation Catheters.
Coronary Dilatation Catheters - Number of participants with Device success (Successful delivery, Successful inflation, Successful deflation, Successful withdrawal) (assessed based on physiological parameters) | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Device success (Successful delivery, Successful inflation, Successful deflation, Successful withdrawal) will be assessed among the patients who receive Coronary Dilatation Catheters. Device success can be summarized as the successful treatment with the device.
Vessel Closure Devices - Number of participants with Composite of access complications | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Composite of access complications (e.g., hematoma, stenosis/occlusion, infection, access site bleeding) will be assessed among the patients who receive Vessel Closure Devices.
Vessel Closure Devices - Number of participants with Successful hemostasis Major and minor bleeding | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Successful hemostasis Major and minor bleeding will be assessed among the patients who receive Vessel Closure Devices.
Vessel Compression Devices - Number of participants with Major and minor bleeding | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Major and minor bleeding will be assessed among the patients who receive Vessel Compression Devices.
Vessel Compression Devices - Number of participants with Complications including: pseudoaneurysm, hematoma (>5cm) in diameter, Hb drop>20 g/L, extended compression time >6 hours, blood transfusion required, bleeding requiring surgical procedure | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Complications including: pseudoaneurysm requiring treatment, hematoma (>5cm) in diameter, Hb drop>20 g/L, extended compression time >6 hours, blood transfusion required, bleeding requiring surgical procedure will be assessed among the patients who receive Vessel Compression Devices.
Vascular Access Introducers - Incidence of safety issues | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Incidence of safety issues (e.g., bleeding, air embolism, hematoma, vessel damage (dissection, perforation, pseudoaneurysm), infection, thrombosis, AV fistula, occlusion, radial artery spasm) will be assessed among the patients who receive Vascular Access Introducers.
Vascular Access Introducers - Incidence of performance issues | During procedure (Start of procedure: defined as time a guidewire first enters the vasculature. End of procedure: defined as vessel closure following the index procedure)
  Incidence of performance issues (e.g., unable to introduce other devices, failure to maintain hemostasis valve integrity, air leakage, bending or kinking of introducer, difficulty inserting/removing the sheath, device breakage detachment or separation, issue with an associated accessory) will be assessed among the patients who receive Vascular Access Introducers.

CONTACTS AND LOCATIONS:
Overall Officials: Chananit Hutson, PhD, Study Director — Abbott Medical Devices
Locations (37):
- United States (7):
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Bryan Heart, Lincoln, Nebraska
  - Ohio State University, Columbus, Ohio
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
- Australia (2):
  - Perth Institute of Vascular Research, Nedlands, WAUS
  - Sir Charles Gairdner Hospital, Nedlands, WAUS
- Universitätsklinik Graz, Graz, Styria, Austria
- Belgium (2):
  - Onze-Lieve-Vrouwziekenhuis Campus Aalst, Aalst, Eflndrs
  - AZ Sint-Blasius Ziekenhuis, Dendermonde, Eflndrs
- China (3):
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jinhua Municipal Central Hospital, Jinhua, Zhejian
  - Ningbo First Hospital, Ningbo, Zhejian
- France (2):
  - CH Chartres, Chartres, Centre-Val de Loire
  - Hôpital Paris Saint-Joseph, Paris, Ile
- Germany (5):
  - Cardioangiologisches Centrum am Bethanien Krankenhaus, Frankfurt am Main, Hesse
  - UNIVERSITATSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz, Rhinela
  - Universitätsklinikum Leipzig AÖR, Leipzig, Saxony
  - Herz- u. Gefäßzentrum Bad Bevensen, Bad Bevensen, Saxon
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schlesw
- Semmelweis University, Budapest, Budapest, Hungary
- Italy (3):
  - Ospedale San Raffaele, Milan, Lombard
  - Centro Cardiologico Monzino, Milan, Lombard
  - Policlinico San Donato, San Donato Milanese, Lombard
- St. Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalon
  - Hospital Universitario de la Paz, Madrid, Madrid
  - Hospital General Universitario de Alicante, Alicante, Valncia
- Switzerland (2):
  - Kantonsspital Aarau, Aarau, Basel
  - Inselspital - University Hospital of Bern, Bern, Canton of Bern
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung, Mtaiwan
  - Cathay General Hospital, Taipei, Ntaiwan
  - National Cheng Kung University Hospital, Tainan, Staiwan
  - Chi Mei Hospital, Tainan, Staiwan
- Al Qassimi Hospital, Sharjah city, Emirate of Sharjah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No